CLINICAL TRIAL: NCT04211246
Title: Efficacy of Oxygen Reserve Index (ORI) to Reduce Hyperoxia in Major Abdominal Surgery
Brief Title: Oxygen Reserve Index to Reduce Hyperoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunah Cho, MD (Other)
Responsible Party: Sponsor-Investigator, Eunah Cho, MD, Clinical Assistant Professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-12-027
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hyperoxemia
MeSH Terms: interventions — Oxygen Saturation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Active Comparator): Fraction of inspired oxygen (FiO2) is titrated guided by SpO2.
  Interventions: Procedure: Titration of fraction of inspired oxygen (FiO2) guided by SpO2
- ORI group (Experimental): Fraction of inspired oxygen (FiO2) is titrated guided by SpO2 and ORI
  Interventions: Procedure: Titration of fraction of inspired oxygen (FiO2) guided by ORI and SpO2

INTERVENTIONS:
Procedure: Titration of fraction of inspired oxygen (FiO2) guided by SpO2 — Titration of fraction of inspired oxygen (FiO2) guided by SpO2
  Other Names: SpO2
  Arms: Standard group
Procedure: Titration of fraction of inspired oxygen (FiO2) guided by ORI and SpO2 — Titration of fraction of inspired oxygen (FiO2) guided by ORI and SpO2
  Other Names: ORI+SpO2
  Arms: ORI group

SUMMARY:
Excessive oxygen administration is known to cause oxidative stress, and absorption atelectasis. Hyperoxia is very common in general anesthesia settings. Even though there are concerns in using excessive oxygen during general anesthesia, the optimal fraction of inspired oxygen (FiO2) for general anesthesia is not well studied.

The oxygen reserve index (ORI) is a parameter which can evaluate partial pressure of oxygen (PaO2) rating from 0 to 1. There are growing evidences in ORI that it might be helpful to reduce hyperoxia in critically ill patients in the intensive care unit, as well as in general anesthesia.

The aim of this study is to evaluate efficacy of oxygen reserve index to reduce hyperoxemia in major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective major abdominal surgery expected to last more than 2hours.
* Patients who are scheduled for invasive arterial cannulation during surgery.

Exclusion Criteria:

* Abnormal pulmonary function test
* Pregnancy
* Saturation of oxygen (SpO2) is below 92% in room air

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Pressure of arterial oxygen (PaO2) after 1 hour of surgery. | After 1 hour of surgery
  Pressure of arterial oxygen is obtain from arterial blood gas analysis as usual practice.

SECONDARY OUTCOMES:
Pressure of arterial oxygen (PaO2) after 2 hours of surgery. | After 2 hours of surgery
  Pressure of arterial oxygen is obtain from arterial blood gas analysis as usual practice.
Pressure of arterial oxygen (PaO2) after 3 hours of surgery. | After 3 hours of surgery
  Pressure of arterial oxygen is obtain from arterial blood gas analysis as usual practice.
Minimal and maximal value of PaO2 throughout the surgery | 1 hour after the end of surgery
  Pressure of arterial oxygen is obtain from arterial blood gas analysis as usual practice.
Fraction of inspired oxygen (FiO2) | 1 hour after the end of surgery
  Fraction of inspired oxygen (FiO2) administered during the surgery
Oxygen reserve index (ORI) | 1 hour after the end of surgery
  Oxygen reserve idex shown from the monitoring device during the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahn JH, Shim JG, Park J, Lee SH, Ryu KH, Cho EA. Oxygen reserve index guided fraction of inspired oxygen titration to reduce hyperoxemia during laparoscopic gastrectomy: A randomized controlled trial. Medicine (Baltimore). 2022 Nov 18;101(46):e31592. doi: 10.1097/MD.0000000000031592. PMID 36401493